CLINICAL TRIAL: NCT00663832
Title: An Open Label, Single Arm, Phase Ib Dose Finding Study of i.v. Panobinostat (LBH589) With Docetaxel and Prednisone in Patients With Hormone Refractory Prostate Cancer
Brief Title: A Dose Finding Study With I.V. Panobinostat (LBH589), Docetaxel, and Prednisone in Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589C2205; 2007-003315-30 (EudraCT Number)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Prostate Cancer
Keywords: Male; Prostate; Cancer; HRPC; DACi
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589 (i.v. panobinostat)

INTERVENTIONS:
Drug: LBH589 (i.v. panobinostat) — i.v. LBH589 dose levels: 10, 15, or 20 mg/m2
  i.v. docetaxel 75 or 60 mg/m2
  oral prednisone 5mg bid.
  LBH589 i.v. administered on days 1 and 8 in combination with docetaxel i.v. on day 1 and prednisone p.o 5mg bid every day of a 21-day cycle
  Other Names: Panobinostat

SUMMARY:
This Phase Ib dose escalation study is designed to characterize the safety, tolerability and preliminary efficacy of i.v. panobinostat (LBH589) in combination with docetaxel and prednisone in the 1st line treatment of patients with hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* HRPC patients
* Evidence of disease progression
* Self care, able to perform light work activities
* Willing to use contraception throughout the study and for 12 weeks after study completion

Exclusion criteria:

* History of other cancers not curatively treated with no evidence of disease for more than 5 years.
* Prior radiotherapy within 3 weeks of starting study treatment
* Prior radiopharmaceuticals (strontium, samarium).
* Impaired cardiac function
* Heart disease
* Liver or renal disease with impaired functions.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of i.v. LBH589 in combination with docetaxel and prednisone in patients with HRPC | determine if MTD occurs after every 3 - 6 pts

SECONDARY OUTCOMES:
To compare the PK profile of i.v. LBH589 with and without docetaxel | PK assessment will occur during the first 2 weeks of each pt treatment. Minor safety throughout the study treatment phase
To determine safety and tolerability of i.v. LBH589 in combination with docetaxel and prednisone in patients with HRPC | PK assessment will occur during the first 2 weeks of each pt treatment
To determine preliminary activity of i.v. LBH589 in combination with docetaxel and prednisone | PK assessment will occur during the first 2 weeks of each pt treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (7):
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Portland, Oregon
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario

REFERENCES:
- See also: Results for CLBH589C2205 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7783